CLINICAL TRIAL: NCT02804802
Title: Impact of DietarY and LIfestyle Risk Factors on Colorectal Cancer Screening (IDYLIC Study). Is it Possible to Target Risk Subjects by Using a Predictive Score?
Brief Title: Impact of DietarY and LIfestyle Risk Factors on Colorectal Cancer Screening
Acronym: IDYLIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRC-K 2011
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire — dietary habits and physical activity questionnaire

SUMMARY:
The main purpose of our project is to construct a lifestyle score based on a short questionnaire easy to complete and to validate it among participants in mass screening for colorectal cancer in Maine and Loire department over the next 2 years (2012 and 2013). We will evaluate the ability of our score to identify subjects with colorectal cancer diagnosed by the screening procedure (Hemoccult II ®, and colonoscopy if the test result is positive). Colorectal cancer will be the primary outcome for the assessment of the score's performance. The secondary endpoint will focus on colorectal adenomas diagnosed by the same procedure. Our secondary objectives are to test a second weighting system, evaluate the benefit in terms of predictive performance to add to the lifestyle score other dietary factors among that have a probable link with the risk of colorectal cancer, determine the acceptability of the questionnaire and to estimate by a cost-utility analysis the impact of applying a strategy of targeted screening using the developed score.

DETAILED DESCRIPTION:
Background: The clinical value of early detection of colorectal cancer has been clearly demonstrated. The evaluation in 23 pilot counties of the organized screening program for colorectal cancer in France, that was widespread throughout the country in 2009, concluded that results are satisfactory but should be improved especially in terms of sensitivity and participation rates. Epidemiological studies show that apart from the hereditary factor and age, the risk of colorectal cancer is mainly associated with lifestyle factors. The World Cancer Research Fund (WCRF) and the American Institute for Cancer Research (AICR) have published jointly in 2007 an update of the scientific knowledge on the relationships between nutritional factors (diet, physical activity) and the risk of cancer. This expert's report confirms that, according to the available data, the risk of colorectal cancer is increased in a convincing way with excessive consumption of alcohol, red meat and processed meat, and among overweight people, especially for those with excess abdominal adiposity. Conversely, the practice of regular physical activity has a protective effect. A recent meta-analysis estimated colorectal cancer relative risks of each of the factors mentioned above, smoking habits and other factors related to lifestyle (obesity, diabetes). This information helps to consider now the development of a predictive score for colorectal cancer.

Objectives: The main purpose of our project is to construct a lifestyle score based on a short questionnaire easy to complete and to validate it among participants in mass screening for colorectal cancer in Maine and Loire department over the next 2 years (2012 and 2013). We will evaluate the ability of our score to identify subjects with colorectal cancer diagnosed by the screening procedure (Hemoccult II ®, and colonoscopy if the test result is positive). Colorectal cancer will be the primary outcome for the assessment of the score's performance. The secondary endpoint will focus on colorectal adenomas diagnosed by the same procedure. Our secondary objectives are to test a second weighting system, evaluate the benefit in terms of predictive performance to add to the lifestyle score other dietary factors among that have a probable link with the risk of colorectal cancer, determine the acceptability of the questionnaire and to estimate by a cost-utility analysis the impact of applying a strategy of targeted screening using the developed score.

Organization: The project will be coordinated by the department of Gastroenterology and Hepatology from Angers University Hospital. All data will be collected at the time of participation in organized screening program for colorectal cancer. The management of data collection will be done in close collaboration with the structure of screening in the Maine et Loire, Cap Santé 49, so as part of a logistic organization that is already operational. The identification of data that are specific to the project will be simplified by using for each participant the same barcode as that for Hemoccult test. To develop a questionnaire adapted to our objectives and a potential future use on large populations, we will rely on the expertise and experience of a French Research Unit in Nutritional Epidemiology (UMR U557 INSERM / INRA / CNAM / Paris XIII University). In recent years, this team has developed scores that assess compliance with the objectives or recommendations of the National Nutrition and Health Program. The Unit also developed a food frequency questionnaire adapted to the French population and has demonstrated the reproducibility and validity of this tool compared to repeated 24 hours dietary records. We will select from this questionnaire the items on the food groups that have an interest with the objectives of this project, our score will be constructed on the basis of consumption of foods or food groups, not nutrients. The statistical analysis will be conducted by the biostatisticians team from Angers University Hospital.

Expected results: The purpose of the tool (the questionnaire and the system for calculating the overall lifestyle score) is to help general practitioners to identify high risk subjects in general population, regardless of familial predisposition, and to encourage these people to participate in the national screening program. Associated with screening based on age, this strategy may optimize colorectal cancer screening in France.

ELIGIBILITY:
Inclusion Criteria:

* All participants in the organized screening for colorectal cancer over the next 2 years in the Maine-et-Loire department.

Exclusion Criteria:

* Personal or family history of polyps or colorectal cancer
* Personal history of bowel disease that already implies a surveillance by colonoscopy (inflammatory bowel syndrome, HNPCC, FAP)
* Diseases with known genetic risk of developing colorectal cancer

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants in the organized screening for colorectal cancer over the next 2 years in the Maine-et-Loire department.
Sampling Method: Non-Probability Sample
Enrollment: 49000 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer diagnosed by colonoscopy after a positive fecal occult blood test (Hemoccult II) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier Caroli-Bosc, MD PhD, Principal Investigator — UH Angers
Locations (1):
- François-Xavier CAROLI-BOSC, Angers, France

IPD SHARING:
Plan to Share IPD: No